CLINICAL TRIAL: NCT06434402
Title: A Virtual, Group-Based, Expressive Writing Intervention for Survivors of Adolescent and Young Adult Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-0440; NCI-2024-04531 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-05-21; First posted 2024-05-30 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Emerging adults (ages18-25 years) (Experimental): Participants complete questionnaires over 20 minutes about their mood, health, and demographic information at baseline, and 1, and 3 months.
  Participants are asked to write about their cancer experiences over 20 minutes (non-stop) for 4 weeks.
  Interventions: Behavioral: Behavioral Intervention
- Young adults (ages 26-39 years) (Experimental): Participants complete questionnaires over 20 minutes about their mood, health, and demographic information at baseline, and 1, and 3 months.
  Participants are asked to write about their cancer experiences over 20 minutes (non-stop) for 4 weeks.
  Interventions: Behavioral: Behavioral Intervention
- General group (ages 18-39 years) (Experimental): Participants complete questionnaires over 20 minutes about their mood, health, and demographic information at baseline, and 1, and 3 months.
  Participants are asked to write about their cancer experiences over 20 minutes (non-stop) for 4 weeks.
  Interventions: Behavioral: Behavioral Intervention

INTERVENTIONS:
Behavioral: Behavioral Intervention — Write about cancer experiences
  Other Names: Behavior Condition Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Treatment

SUMMARY:
To learn more about the experiences of adolescent and young adult cancer survivors and investigate whether a group-based writing intervention can help to improve quality of life of adolescent and young adult cancer survivors.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the feasibility of a virtual, group-based expressive writing intervention for survivors of adolescent and young adult cancer.

Secondary Objective:

To preliminarily assess the impact of the study for cancer survivors.

ELIGIBILITY:
Inclusion criteria:

* Age 15 - 39 years at cancer diagnosis
* Age 18 - 39 years at study entry
* Diagnosed between 1 and 5 years ago prior to enrollment
* Can speak, read, and write in English

Exclusion criteria:

* Nonmelanoma skin cancer
* Major mental health disorder (e.g., schizophrenia or bipolar disorder [determined from patient records or self-disclosure])
* No internet access.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Study Completion Rate | At 1 month follow-up
  The Study completion rate is defined as the average proportion of participants who complete follow-up assessments at 1-month follow-up. We will also calculate the 95% confidence intervals for the study completion rate.
Intervention Adherence Rate | At the end of intervention (week 8)
  The intervention adherence rate will be calculated as the number of completed writing tasks divided by the total number of assigned tasks (4).

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy-General | Baseline, and 1- and 3-month follow-up
  The Functional Assessment of Cancer Therapy-General will be used to measure multidimensional quality of life, encompassing physical, social, emotional, and functional well-being, across 27 items. Each item is rated on a 5-point Likert scale ranging from 0 to 4. The overall score can range from 0 to 108, with higher scores indicating a better quality of life.
Perceived Stress | Baseline, and 1- and 3-month follow-up
  The Perceived Stress scale will be used to measure perceived stress. This 4-item measure assesses the degree to which situations in one's life are appraised as stressful. The overall score can range from 0 to 16, with higher scores indicating higher perceived stress.
Coping self-efficacy | Baseline, and 1- and 3-month follow-up
  The Cancer Behavior Inventory will be used to measure self-efficacy for coping with cancer. Each item is rated on a 9-point Likert scale. The total score ranges from 9 to 81, with higher scores indicating greater self-efficacy for coping with cancer.
Impact of Event Scale | Baseline, and 1- and 3-month follow-up
  The 5-item intrusion subscale of the Impact of Event Scale will be used to assess unwanted thoughts related to cancer. Each item is rated on a 4-point Likert scale. The total score ranges from 0 to 25, with higher scores indicating a greater frequency and intensity of intrusive thoughts.
Common Humanity & Self-Kindness | Baseline, and 1- and 3-month follow-up
  Common Humanity and Self-Kindness will be measured using the subscales of the Self-Compassion Scale. These subscales capture positive aspects of self-compassion, including self-kindness (e.g., "When I am going through a very hard time, I give myself the caring and tenderness I need") and common humanity (e.g., "When I am down and out, I remind myself that there are lots of other people in the world feeling like me"). Each item is rated on a 5-point Likert scale. The total score for each subscale ranges from 5 to 25, with higher scores indicating a stronger sense of common humanity and self-kindness.
Posttraumatic growth | Baseline, and 1- and 3-month follow-up
  The Posttraumatic Growth Inventory will be used to assess perceived positive changes as a result of a specific traumatic event. It includes 9 items, each rated on a 6-point Likert scale. The total score ranges from 0 to 45, with higher scores indicating greater perceived posttraumatic growth.

CONTACTS AND LOCATIONS:
Overall Officials: Qian Lu, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org